CLINICAL TRIAL: NCT06132451
Title: In-Hospital Detection of Elevated Blood Pressure (INDEBP): Prevalence of New or Uncontrolled Hypertension and Safety of Postponement of Antihypertensive Treatment Adaption in Medical In-patients
Brief Title: In-Hospital Detection of Elevated Blood Pressure
Acronym: INDEBP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Annina Vischer (Other)
Responsible Party: Sponsor-Investigator, Annina Vischer, Principle Investigator, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: INDEBP-prospective; 2023-01566 (Other: EKNZ)
Record Dates: First submitted 2023-11-05; First posted 2023-11-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hypertension; Blood Pressure, High
Keywords: arterial hypertension; elevated blood pressure; ambulatory blood pressure measurement; antihypertensive medication
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: There will be block-wise randomization. During the first block, the study team will not interfere with the treating physician, in order to ensure that they will treat the patient according to what they perceive as the current usual practice. During the second block the patients receive no change of their original antihypertensive treatment.
Who Masked: Care Provider
Masking Description: In the first block, the treating physicians will not be informed about the study participation of their patient, in order to ensure that they will treat the patient according to what they perceive as the current usual practice. In the second block, the treating physicians will be informed about the study participation of their patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual practice arm (No Intervention): Patients will be treated according to their treating physicians' decision.
- Postponement of treatment arm (Other): Antihypertensive treatment adaptions will be postponed until after a 24h ambulatory blood pressure measurement (ABPM) 4 weeks after hospital discharge.
  Interventions: Other: Postponement of antihypertensive treatment

INTERVENTIONS:
Other: Postponement of antihypertensive treatment — Hypertensive blood pressure values in medical in-patients will not be treated during hospitalisation until confirmed by ABPM 4 weeks after hospital discharge
  Arms: Postponement of treatment arm

SUMMARY:
The goal of this clinical trial is to analyse the prevalence of new or uncontrolled arterial hypertension (AHT) after hospital discharge of medical in-patients with elevated blood pressure (BP) values during hospitalisation.

The main questions it aims to answer are:

* Do elevated BP values during hospitalisation correspond to new or uncontrolled AHT after hospital discharge?
* Is it safe to postpone adaption of antihypertensive treatment until after proper evaluation of AHT after hospital discharge?

Participants will either be treated according to their physicians' decision or antihypertensive treatment adaptions will be postponed until after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized on the internal medicine ward for non-cardiovascular causes, i.e. patients hospitalized for conditions, which are not acutely worsened by uncontrolled AHT
* Asymptomatic elevated BP values (defined as 140-180 mmHg systolic and/or 90-110 mmHg diastolic) on at least 2 occasions
* Ability to understand study procedures and to provide written informed consent

Exclusion Criteria:

* Hospitalization for any conditions which can be worsened by uncontrolled AHT:
* Cerebrovascular events
* Acute coronary syndrome
* Acute or decompensated heart failure
* Any condition preventing ABPM
* Pregnant or lactating women
* Failure to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of persisting new or uncontrolled arterial hypertension | 4 weeks after hospital discharge
  Elevated blood pressure values in ambulatory blood pressure monitoring
Prevalence of a combined hypertensive complication endpoint | Until 4 weeks after hospital discharge
  Consisting of intracerebral bleeding, ischemic stroke, myocardial infarction, cardiovascular death or cardiovascular re-hospitalization
Prevalence of a combined hypotensive complication endpoint | Until 4 weeks after hospital discharge
  Consisting of falls, acute kidney injury, electrolyte disturbances, re-hospitalizations due to hypotension, or BP values on ABPM below the lower treatment limit

SECONDARY OUTCOMES:
Clinic blood pressure measurement in mmHg | At baseline
  Documented in the patient documentation
Research blood pressure measurement in mmHg | At baseline
  Standardized blood pressure measurement taken by research staff
Prevalence of previously unknown arterial hypertension | At baseline
  No previously documented diagnosis of arterial hypertension and no antihypertensive treatment
Prevalence of female gender | At baseline
  As reported by participant
Prevalence of re-hospitalization for any cause | Until 4 weeks after hospital discharge
  According to hospital documentation and patient interrogation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No